CLINICAL TRIAL: NCT00770419
Title: Perception of Caregiver Burden
Brief Title: Perceptions of Burden in Patients With Late-Stage Cancer and Their Caregivers
Status: Withdrawn | Type: Observational
Why Stopped: Slow accrual
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Rutgers Cancer Institute of New Jersey (Other)
Responsible Party: Sponsor
Other Study IDs: 130601; P30CA072720 (NIH); CDR0000597594; CINJ-IRB-0220080083
Record Dates: First submitted 2008-10-09; First posted 2008-10-10 (Estimated); Last update posted 2015-05-29 (Estimated); Status verified 2015-05

CONDITIONS: Brain and Central Nervous System Tumors; Chronic Myeloproliferative Disorders; Depression; Leukemia; Lymphoma; Multiple Myeloma and Plasma Cell Neoplasm; Myelodysplastic Syndromes; Myelodysplastic/Myeloproliferative Neoplasms; Psychosocial Effects of Cancer and Its Treatment; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: depression; psychosocial effects of cancer and its treatment; unspecified adult solid tumor, protocol specific; acute undifferentiated leukemia; adult acute lymphoblastic leukemia in remission; adult acute myeloid leukemia in remission; adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with t(15;17)(q22;q12); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with t(8;21)(q22;q22); atypical chronic myeloid leukemia, BCR-ABL negative; chronic myelomonocytic leukemia; mast cell leukemia; meningeal chronic myelogenous leukemia; prolymphocytic leukemia; recurrent adult acute lymphoblastic leukemia; recurrent adult acute myeloid leukemia; recurrent adult T-cell leukemia/lymphoma; refractory chronic lymphocytic leukemia; refractory hairy cell leukemia; relapsing chronic myelogenous leukemia; secondary acute myeloid leukemia; T-cell large granular lymphocyte leukemia; AIDS-related diffuse large cell lymphoma; AIDS-related diffuse mixed cell lymphoma; AIDS-related diffuse small cleaved cell lymphoma; AIDS-related immunoblastic large cell lymphoma; AIDS-related lymphoblastic lymphoma; AIDS-related peripheral/systemic lymphoma; AIDS-related primary CNS lymphoma; AIDS-related small noncleaved cell lymphoma; HIV-associated Hodgkin lymphoma; recurrent adult Hodgkin lymphoma; anaplastic large cell lymphoma; angioimmunoblastic T-cell lymphoma; cutaneous B-cell non-Hodgkin lymphoma; recurrent cutaneous T-cell non-Hodgkin lymphoma; recurrent mycosis fungoides/Sezary syndrome; adult grade III lymphomatoid granulomatosis; adult nasal type extranodal NK/T-cell lymphoma; Waldenstrom macroglobulinemia; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma; recurrent adult Burkitt lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult grade III lymphomatoid granulomatosis; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent mantle cell lymphoma; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; intraocular lymphoma; primary central nervous system non-Hodgkin lymphoma; primary central nervous system Hodgkin lymphoma; chronic eosinophilic leukemia; chronic neutrophilic leukemia; primary myelofibrosis; primary systemic amyloidosis; refractory multiple myeloma; previously treated myelodysplastic syndromes; secondary myelodysplastic syndromes; myelodysplastic/myeloproliferative neoplasm, unclassifiable
MeSH Terms: conditions — Central Nervous System Neoplasms; Myeloproliferative Disorders; Depression; Leukemia; Lymphoma; Multiple Myeloma; Neoplasms, Plasma Cell; Myelodysplastic Syndromes; Myelodysplastic-Myeloproliferative Diseases; Leukemia, Biphenotypic, Acute; Congenital Abnormalities; Leukemia, Myeloid, Chronic, Atypical, BCR-ABL Negative; Leukemia, Myelomonocytic, Chronic; Leukemia, Mast-Cell; Leukemia, Prolymphocytic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Hairy Cell; Leukemia, Large Granular Lymphocytic; Hodgkin Disease; Lymphoma, Large-Cell, Anaplastic; Immunoblastic Lymphadenopathy; Lymphoma, T-Cell, Cutaneous; Mycosis Fungoides; Sezary Syndrome; Lymphoma, Extranodal NK-T-Cell; Waldenstrom Macroglobulinemia; Lymphoma, B-Cell, Marginal Zone; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Lymphoma, Large-Cell, Immunoblastic; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Intraocular Lymphoma; Pdgfra-Associated Chronic Eosinophilic Leukemia; Leukemia, Neutrophilic, Chronic; Primary Myelofibrosis; Immunoglobulin Light-chain Amyloidosis | interventions — Psychiatric Rehabilitation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: medical chart review
Other: questionnaire administration
Procedure: psychosocial assessment and care

SUMMARY:
RATIONALE: Gathering information over time about patients' sense of being a burden on their caregiver, and caregivers' sense of burden on themselves, may help doctors learn more about the desire to die in patients with late-stage cancer.

PURPOSE: This clinical trial is studying perceptions of burden in patients with late-stage cancer and their caregivers.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To measure psychosocial correlates of desire for hastened death (DHD) and change in DHD in patients with late-stage cancer by examining the relationship among a patient's perception of being a burden, their caregiver's perceptions of the patient's burdensomeness, and DHD changes over time.

Secondary

* To identify coping and personality factors in both caregivers and patients that may be related to the patients' DHD and changes in their DHD.

OUTLINE: Patients and caregiver dyads complete questionnaires at baseline, 2 months, and 4 months. The dyads complete demographic questionnaire, the Hospital Anxiety and Depression Scale (HADS), the Beck Hopelessness Scale (BHS), the Dyadic Adjustment Scale (DAS), and the Life Orientation Test-Revised (LOT-R). Patients also complete the Schedule of Attitudes Toward Hastened Death (SAHD), the Brief Coping Orientation to Problems Experienced (Brief COPE), the Memorial Symptom Assessment Scale-Short Form (MSAS-SF), and the Caregiver Demands Scale (CDS). Caregivers also complete the Katz Index of Independence in Activities of Daily Living (IADL).

Patients' medical charts are reviewed for stage and node status at primary diagnosis, previous oncology surgeries, previous adjuvant treatments, treatment at time of recurrence, disease free interval, site of metastasis, and response to current treatment.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Meets 1 of the following criteria

  * Patient with a diagnosis of cancer

    * Confirmed late-stage disease refractory to standard primary therapy
    * Reside with a non-paid primary caregiver
    * Receiving care at the Cancer Institute of New Jersey
  * Caregiver

    * Must be at least 18 years old

PATIENT CHARACTERISTICS:

* Life expectancy ≥ 4 months
* No documented or observable cognitive (e.g., dementia) or psychiatric (e.g., psychosis) problems that would interfere with study participation
* Able to read and write English (patient and caregiver)

PRIOR CONCURRENT THERAPY:

* Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Caregivers and patients with late-stage oncological disease.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2008-05; Primary Completion 2010-01 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Relationship between patient's sense of being a burden on primary caregiver & increase in patient desire for hastened death (DHD) by Caregiver Demands Scale (CDS) at baseline & Schedule of Attitudes toward Hastened Death (SAHD) at 2 & 4 mo.
Contribution of the caregiver's sense of caregiver burden, as measured by the caregiver version of the CDS at baseline, on increases in patient DHD over time

SECONDARY OUTCOMES:
Identification of coping and personality factors in both caregivers and patients that may be related to the patients' DHD and changes in their DHD

CONTACTS AND LOCATIONS:
Overall Officials: Linda Patrick-Miller, PhD, Principal Investigator — Rutgers Cancer Institute of New Jersey